CLINICAL TRIAL: NCT03230851
Title: the Efficacy and Safety of Indobufen and Low-dose Aspirin in Different Regimens of Antiplatelet Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 006
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Coronary Atherosclerosis
Keywords: Light Transmittance Aggregometry; Indobufen; Aspirin; Plasma Thromboxane; Urine 11-dehydro thromboxane
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Therapeutics; indobufen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- aspirin 100mg/d therapy (Experimental): Group1: aspirin 100 mg/d;
  Interventions: Drug: aspirin 100mg/d therapy
- aspirin 100mg/2d therapy (Experimental): Group2: aspirin ;
  Interventions: Drug: aspirin 100mg/2d therapy
- aspirin 100mg/3d therapy (Experimental): Groups3: aspirin ;
  Interventions: Drug: aspirin 100mg/3d therapy
- aspirin 50mg bid therapy (Experimental): Groups4: morning 50mg evening 50mg;
  Interventions: Drug: aspirin 50mg bid therapy
- aspirin 75mg/d therapy (Experimental): Group5: aspirin 75mg / d;
  Interventions: Drug: aspirin 75mg/d therapy
- aspirin 50mg/d therapy (Experimental): Group6: aspirin 50mg / d;
  Interventions: Drug: aspirin 50mg/d therapy
- indobufen 100mg bid therapy (Experimental): Group7: 100mg bid
  Interventions: Drug: indobufen 100mg bid therapy

INTERVENTIONS:
Drug: aspirin 100mg/d therapy — 100mg aspirin for at least 5 days followed by aspirin 100mg/d
  Arms: aspirin 100mg/d therapy
Drug: aspirin 100mg/2d therapy — 100mg aspirin for at least 5 days followed by aspirin 100mg/2d
  Arms: aspirin 100mg/2d therapy
Drug: aspirin 100mg/3d therapy — 100mg aspirin for at least 5 days followed by aspirin 100mg/3d
  Arms: aspirin 100mg/3d therapy
Drug: aspirin 50mg bid therapy — 100mg aspirin for at least 5 days followed by aspirin 50mg bid
  Arms: aspirin 50mg bid therapy
Drug: aspirin 75mg/d therapy — 100mg aspirin for at least 5 days followed by aspirin 75mg/d
  Arms: aspirin 75mg/d therapy
Drug: aspirin 50mg/d therapy — 100mg aspirin for at least 5 days followed by aspirin 50mg/d
  Arms: aspirin 50mg/d therapy
Drug: indobufen 100mg bid therapy — 100mg aspirin for at least 5 days followed by indobufen 100mg bid
  Arms: indobufen 100mg bid therapy

SUMMARY:
A total of 210 coronary atherosclerosis patients without indications for stent implantation are included. The baseline values of platelet aggregation rate, plasmaThromboxaneB2 and urinary 11-dh ThromboxaneB2 are measured by Light Transmittance Aggregometry method and ELISA after aspirin 100 mg /d ≥5d. Then the patients are randomly divided into 7 groups: Group1: aspirin 100 mg/d; Group2: aspirin 100 mg /2d; Groups3: aspirin 100 mg / 3d; Groups4: morning 50mg evening 50mg; Group5: aspirin 75mg / d; Group6: aspirin 50mg / d; Group7: indobufen100mg bid. One month later,arachidonic acid-induced platelet aggregation rate , plasma TXB2 and urine 11-dh TXB2 are analyzed again. All patients are followed-up for 1 year. The stomach Intestinal reactions, small bleeding events are recorded.

DETAILED DESCRIPTION:
A total of 210 coronary atherosclerosis patients without indications for stent implantation are included. Exclusion criteria：Aspirin resistance, uncontrolled hypertension (> 160 / 100mmHg),hemoglobin concentration <100g /L, hemorrhagic disease or a history of bleeding tendency, taking other nonsteroidal drugs, severe liver disease history, malignant tumor, active gastric mucosa bleeding, percutaneous coronary intervention history, coronary artery bypass surgery, cardiac function grade Ⅳ.The baseline values of platelet aggregation rate, plasma TXB2 and urinary 11-dh TXB2 are measured by LTA method and ELISA after aspirin 100 mg /d ≥5d. Then the patients are randomly divided into 7 groups: Group1: aspirin 100 mg/d; Group2: aspirin 100 mg /2d; Groups3: aspirin 100 mg / 3d; Groups4: morning 50mg evening 50mg; Group5: aspirin 75mg / d; Group6: aspirin 50mg / d; Group7: indobufen100mg bid. One month later,arachidonic acid-induced platelet aggregation rate , plasma TXB2 and urine 11-dh TXB2 are analyzed again. All patients are followed-up for 1month,6months and1 year. The stomach Intestinal reactions, small bleeding events ,whether to take proton pump inhibitors are recorded.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of coronary atherosclerosis without indications for stent implantation .

Patient aged >18 years and ≤75years. Must be able to swallow tablets

Exclusion Criteria:

Aspirin resistance; uncontrolled hypertension (> 160 / 100mmHg); hemoglobin <100g / L; hemorrhagic disease or bleeding tendency history; taking other non-steroidal drugs; severe liver disease history; malignant neoplasms; active gastric mucosa bleeding; PCI history; coronary artery bypass surgery; cardiac function grade Ⅳ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-08-20 (Estimated); Primary Completion 2018-07-10 (Estimated); Study Completion 2018-08-10 (Estimated)

PRIMARY OUTCOMES:
platelet aggregation | 2 hours
  Regional differences between blood samples from each subjects of different groups by LTA.The results of LTA are reported in platelet aggregation rate(%).Platelet aggregation was induced by0.5mg/ml arachidonic acid (AA).
plasma thromboxaneB2 | 3montshs
  The plasma thromboxane B2 concentration of each subjects are measured by enzyme-linked immunosorbent assay .(cayman chemical, thromboxaneB2 express EIA kit-Monoclonal)
urine 11-dehydro thromboxaneB2 | 3 months
  The urine 11-dehydro thromboxane B2 concentration of each subjects are measured by ELISA.(cayman chemical,11-dehydro thromboxaneB2 ELISA kit-Monoclonal)

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China